CLINICAL TRIAL: NCT01218581
Title: Aromatase Inhibitors or Gonadotropin-releasing Hormone Agonists for the Management of Uterine Adenomyosis: A Randomized Controlled Trial
Brief Title: Aromatase Inhibitors or GnRH-a for Uterine Adenomyosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Prof. Ahmed Badawy, Mansoura Faculty of Medicine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: adenomyosis; aromatase inhibitors
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Last update posted 2010-10-11 (Estimated); Status verified 2005-12

CONDITIONS: the Efficacy of Aromatase Inhibitor vs. Gonadotrpins Releasing Hormone Agonists in Treating Premenopausal Women With Uterine Adenomyosis
Keywords: Adenomyosis, letrozole, GnRH-a
MeSH Terms: conditions — Adenomyosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group A (Active Comparator): Group A received oral letrozole (2.5 mg/day, Femara, Novartis PharmaServices, Basel, Switzerland)
  Interventions: Drug: received oral letrozole (2.5 mg/day)and goserelin subcutaneosly (3.6 mg/month)
- group B (Active Comparator): group B received goserelin subcutaneosly (3.6 mg/month, Zoladex@, Zeneka Pharma International, UK)
  Interventions: Drug: received oral letrozole (2.5 mg/day)and goserelin subcutaneosly (3.6 mg/month)

INTERVENTIONS:
Drug: received oral letrozole (2.5 mg/day)and goserelin subcutaneosly (3.6 mg/month)

SUMMARY:
To date, there is no uniform agreement on the most appropriate therapeutic methods for managing women with uterine adenomyosis and/or adenomyoma who want to preserve their fertility. Management with hormonal treatment that aims to reduce the proliferation of endometrial cells is promising, but there is a paucity of well-designed studies to guide treatment. There is a strong need to develop pharmacological agents that provide an efficient outcome. Gonadotripn releasing hormone analogues (GnRHa) have been used in several studies, to produce a constant hypoestrogenic state in a woman with adenomyosis which cause amenorrhoea, control of pain and uterine shrinkage . Pure antiestrogens, however, may offer some advantage in the treatment of adenomyosis and trials are required to assess its usefulness. Leiomyoma and uterine volumes were successfully reduced by use of aromatase inhibitors (AIs). Assuming aromatase production activity in the adenomyosis lesion, Kimura et al, used GnRHa and an AI concomitantly for treatment of uterine adenomyosis. This lack of information stimulated us to run this trial to compare the efficacy of aromatase inhibitor vs. GnRHa in treating premenopausal women with uterine adenomyosis.

DETAILED DESCRIPTION:
This is a prospective, randomized, non-blind trial performed in the period from December 2005 and January 2010 in the teaching hospitals affiliated with Mansoura University (Egypt) and a private practice setting (Delta Fertility Center, Egypt). Thirty eight patients were assessed for eligibility, 6 patients were excluded and 32 with uterine adenomyosis were included in the study. Patients included in the study were premenopausal women aged 18-42 years with adenomyosis with abnormal uterine bleeding, unexplained infertility, pelvic pain, dysmenorrhea, or pressure effect. Excluded subjects included women who had myoma(s) measuring >2 cm, women with uterine adenomyoma who were under treatment with any type of hormonal therapy more recently than 1 month, and women with a history of major medical problem and/or previous medical or surgical treatment for the problem.

Patients were randomly allocated into two treatments groups (A and B) using a computer-generated random table. Group A received oral letrozole (2.5 mg/day, Femara, Novartis PharmaServices, Basel, Switzerland) and group B received goserelin subcutaneosly (3.6 mg/month, Zoladex@, Zeneka Pharma International, UK) for 12 weeks. Because, for technical reasons, GnRHa was supplied in vials and aromatase inhibitor in tablets, a double-blind study design was not feasible. Instead an assessor-blind design was chosen, whereby preparation and administration were performed by a person who did not take part in any decision concerning medication administration during the study. The study was approved by the ethics committee of the university and institutional Review Board (IRB), and each subject provided written informed consent before participating in the study. All subjects underwent baseline measurement, performed in the early follicular phase.

An expert gynecologist performed all transvaginal ultrasound scans and analysis using D 4000 (Honda, Japan) ultrasound machine with a 5.5-MHz vaginal probe. Ultrasound criteria used for diagnosis of adenomyosis included uterine enlargement in the absence of leiomyomas, asymmetric enlargement of the anterior or posterior myometrial wall, lack of contour abnormality or mass effect, heterogeneous, poorly circumcised areas within the myometrium, hyperechoic islands or nodules, finger-like projections or linear striations. After identification of the adenomyosis, its volume was calculated with a stepwise planimetry method using an integrated software program. Measurements for the whole uterine and the adenomyoma volumes were performed at baseline and during treatment at weeks 4, 8, and 12. Symptoms at the start and after 12 weeks of therapy were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the study were premenopausal women aged 18-42 years with adenomyosis with abnormal uterine bleeding, unexplained infertility, pelvic pain, dysmenorrhea, or pressure effect

Exclusion Criteria:

* Excluded subjects included women who had myoma(s) measuring >2 cm, women with uterine adenomyoma who were under treatment with any type of hormonal therapy more recently than 1 month, and women with a history of major medical problem and/or previous medical or surgical treatment for the problem

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate, Egypt